CLINICAL TRIAL: NCT01318382
Title: Residual Curarization and Its Incidence at Tracheal Extubation
Brief Title: Residual Curarization and Its Incidence at Tracheal Extubation (P08194)
Acronym: RECITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P08194; MK-8616-063 (Other: Merck Protocol ID)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Observation of Neuromuscular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TOF-Watch SX® (Experimental): Participants who have undergone elective open or laparoscopic abdominal surgery, received general anesthesia, received at least one dose of non-depolarizing neuromuscular blocker and had the extent of their recovery from NMB monitored by a TOF-Watch SX®.
  Interventions: Device: TOF-Watch SX® Monitoring of NMB

INTERVENTIONS:
Device: TOF-Watch SX® Monitoring of NMB — Participants will have the extent of NMB monitored by a TOF-Watch SX®.

SUMMARY:
This study will assess the residual neuromuscular blockade (NMB) Train-Of-Four (TOF) ratios at tracheal extubation when anesthesiologists have determined that full recovery of neuromuscular function has occurred using standard clinical criteria for participants whose non-depolarizing-induced NMB is either not reversed or reversed with an acetylcholinesterase inhibitor administered as per standard routine care.

DETAILED DESCRIPTION:
This is an observational cohort study with a device intervention to determine in which cohort the subject is falling.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be American Society of Anesthesia (ASA) class 1-3.
* Participant must be scheduled for elective open or laparoscopic abdominal surgery that is anticipated to last less than 4 hours.
* Administration of general anesthesia and ≥ 1 dose of non-depolarizing neuromuscular blockers for endotracheal intubation or maintenance of neuromuscular blockade.
* Extubation must occur in the operating room (OR).

Exclusion Criteria:

* Surgery re-admission on the same hospital admission.
* Pre-established need for or expected to require post-operative mechanical ventilation.
* Conditions, surgical procedures or position that may interfere with the TOF-Watch SX® operation, calibration or accuracy.
* Administration of sugammadex (Bridion®) for reversal of neuromuscular blockade.
* Participation in any other clinical trial.
* Member or a family member of the personnel of the investigational or Sponsor staff directly involved with this trial.
* Anesthesiologist use of objective neuromuscular monitoring during surgery (e.g. mechanomyography, electromyography or related method).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

REFERENCES:
- [Result] Fortier LP, McKeen D, Turner K, de Medicis E, Warriner B, Jones PM, Chaput A, Pouliot JF, Galarneau A. The RECITE Study: A Canadian Prospective, Multicenter Study of the Incidence and Severity of Residual Neuromuscular Blockade. Anesth Analg. 2015 Aug;121(2):366-72. doi: 10.1213/ANE.0000000000000757. PMID 25902322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 8 sites in Canada between June 2011 and May 2012.
Groups:
- TOF-Watch SX®: All enrolled participants who had undergone elective open or laparoscopic abdominal surgery, received general anesthesia, received at least one dose of non-depolarizing neuromuscular blocker and had the extent of their recovery from neuromuscular blockade (NMB) monitored by a TOF-Watch SX®.
Period: Overall Study
Arm/Group | TOF-Watch SX®
Started | 302
Completed | 289
Not Completed | 13
Not completed — Physician Decision | 2
Not completed — Device Malfunction | 10
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- TOF-Watch SX®: All enrolled participants who had undergone elective open or laparoscopic abdominal surgery, received general anesthesia, received at least one dose of non-depolarizing neuromuscular blocker and had the extent of their recovery from NMB monitored by a TOF-Watch SX®.
Arm/Group | TOF-Watch SX®
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222
  Male | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Residual Neuromuscular Blockade (NMB)(Train of Four [TOF] Ratio <0.9) at Time of Tracheal Extubation
Description: Neuromuscular functioning was monitored at time of tracheal extubation by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB. A T4/T1 Ratio of <0.9 is indicative of residual NMB.
Time Frame: Up to 1 minute prior to tracheal extubation
Population: Per-Protocol Population was defined as all enrolled participants for whom TOF-Watch SX® measurements were collected and had an evaluable TOF Ratio at time of tracheal extubation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- TOF-Watch SX®: All enrolled participants who had undergone elective open or laparoscopic abdominal surgery, received general anesthesia, received at least one dose of non-depolarizing neuromuscular blocker, had the extent of their recovery from NMB monitored by a TOF-Watch SX® and had an evaluable TOF Ratio at time of tracheal extubation.
Arm/Group | TOF-Watch SX®
Number analyzed (Participants) | 241
percentage of participants | 56 [49.7 to 62.3]

2. Secondary Outcome: Percentage of Participants With Residual NMB (TOF Ratio <0.9) Upon Arrival to the Post-anesthesia Care Unit (PACU)
Description: Neuromuscular functioning was monitored at time of PACU arrival by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB. A T4/T1 Ratio of <0.9 is indicative of residual NMB.
Time Frame: Up to 2 minutes prior to PACU arrival
Population: The PACU Population was defined as all enrolled participants for whom TOF-Watch SX® measurements were collected and had an evaluable TOF Ratio at time of PACU arrival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- TOF-Watch SX®: All enrolled participants who had undergone elective open or laparoscopic abdominal surgery, received general anesthesia, received at least one dose of non-depolarizing neuromuscular blocker, had the extent of their recovery from NMB monitored by a TOF-Watch SX® and had an evaluable TOF Ratio at time of PACU arrival.
Arm/Group | TOF-Watch SX®
Number analyzed (Participants) | 207
percentage of participants | 44 [37.7 to 50.2]

3. Secondary Outcome: Percentage of Participants With Residual NMB at Various TOF Ratios (<0.6, ≥0.6 to <0.7, ≥0.7 to <0.8, ≥0.8 to <0.9) at Tracheal Extubation
Description: Neuromuscular functioning was monitored at time of tracheal extubation by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB.
Time Frame: Up to 1 minute prior to tracheal extubation
Population: The Per-Protocol Population was defined as all enrolled participants for whom TOF-Watch SX® measurements were collected and had an evaluable TOF Ratio at time of tracheal extubation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOF-Watch SX®
Number analyzed (Participants) | 241
percentage of participants
  TOF Ratio <0.6 | 19.1 [14.1 to 24.0]
  TOF Ratio ≥0.6 to <0.7 | 11.6 [7.6 to 15.7]
  TOF Ratio ≥0.7 to <0.8 | 8.7 [5.2 to 12.3]
  TOF Ratio ≥0.8 to <0.9 | 16.6 [11.9 to 21.3]
  TOF Ratio ≥0.9 | 44.0 [37.7 to 50.3]

4. Secondary Outcome: Percentage of Participants With Residual NMB at Various TOF Ratios (<0.6, ≥ 0.6 to <0.7, ≥ 0.7 to <0.8, ≥0.8 to <0.9) Upon Arrival to the PACU
Description: Neuromuscular functioning was monitored at time of PACU arrival by applying three TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB.
Time Frame: Up to 2 minutes prior to PACU arrival
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TOF-Watch SX®
Number analyzed (Participants) | 207
percentage of participants
  TOF Ratio <0.6 | 7.7 [4.4 to 11.1]
  TOF Ratio ≥0.6 to <0.7 | 7.2 [4.0 to 10.5]
  TOF Ratio ≥0.7 to <0.8 | 13.5 [9.2 to 17.8]
  TOF Ratio ≥0.8 to <0.9 | 15.5 [10.9 to 20.0]
  TOF Ratio ≥0.9 | 56.0 [49.8 to 62.3]

ADVERSE EVENTS:
Time Frame: Through Day 1 (up to one day after surgery)
Description: The All Enrolled Participants population consisted of all participants meeting eligibility criteria who were enrolled into the study.
Arm/Group | TOF-Watch SX®
Serious Adverse Events (participants affected / at risk) | 24/302
Other Adverse Events (participants affected / at risk) | 0/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOF-Watch SX® (N=302)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Clostridial Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Anastomotic Leak (Injury, poisoning and procedural complications) | 2 (2)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram T Wave Inversion (Investigations) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 3 (3)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Explorative Laparotomy (Surgical and medical procedures) | 1 (1)
Hypovolaemic Shock (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide copies of abstracts or manuscripts for publication that report any results of the trial to the Sponsor 45 days prior to submission for publication or presentation.